CLINICAL TRIAL: NCT01475201
Title: Step Monitoring to Improve ARTERial Health
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Associate Professor of Medicine and Physician Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR-MOP-114996
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: Type 2 diabetes; Hypertension; Primary Care; Physical Activity; Behavioural Intervention; Pedometer; Accelerometer; Arterial Stiffness; Carotid femoral pulse wave velocity; Vascular disease risk; Vascular disease prevention; Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Step Count Prescription Arm (Experimental): The active trial arm intervention consists of usual care plus step count prescription delivered by the treating doctor, over a one-year period.
  Interventions: Behavioral: Step count prescription
- Usual care arm (Active Comparator): The control trial arm will receive usual care alone, over a one-year period (i.e. no step count prescription but, in accordance with guidelines, including advice to engage in 30-60 minutes of activity on most days of the week). Consistent with clinical practice guidelines, our collaborating doctors have indicated that the usual care of the target population requires clinic visits at roughly three-month intervals to ensure vascular risk factor monitoring and management.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Step count prescription — Treating physicians will provide a pedometer, pedometer log, and step count prescription. The aim is a net increase of at least 3,000 steps/day over one year. The time frame for this increase will be 10 months for sedentary participants (<5,000 steps/day), 7 months for low active participants (5,000-7,499 steps/day), and 5 months for somewhat active participants (7,500-9,999 steps/day). If goals are not met, the doctor and participant will review barriers and facilitators, and a more individualized prescription will be formulated (e.g. lower incremental step count targets or slower rate of dose escalation). For participants who meet goals, the doctor and participant will together decide whether to aim for a further increase.
  Arms: Step Count Prescription Arm
Behavioral: Usual care — The control trial arm will receive usual care alone, over a one-year period (i.e. no step count prescription but, in accordance with guidelines, including advice to engage in 30-60 minutes of activity on most days of the week).
  Arms: Usual care arm

SUMMARY:
Many people with diabetes and/or high blood pressure (hypertension) are not very active. When people are more active, they can reduce the chances of having a heart attack or stroke. Walking more is a cheap and effective way to be more active and to lower the risk of heart attacks and strokes. The problem is that many people do not walk enough! The investigators will study if people with diabetes and/or hypertension walk more when the doctor gives them a prescription with the number of steps they should be walking every day. The investigators will compare this group, called 'active', to another group, called 'control', in which doctors and their patients do what they usually do, over a period of one year.

The investigators will measure the number of steps the investigators walk everyday with a step counter or pedometer. In the step count prescription group, the doctors will give to the 'active' group a pedometer, a step count record book, and step count prescriptions. The overall goal is to gradually increase daily steps. The speed of the increase in step count will be slower for less active people. At each visit the doctor will look at the step count record book. The doctor will then give a new step count prescription to the patients. Patients of the two groups will see their doctor about four times during the year, which is how often they usually see their doctor. At the end of one year, the investigators will see the difference in the hardness of the arteries between the 'active' and the 'control' groups, using simple and safe measurements, similar to ultrasound in pregnant ladies. People with hard arteries are more likely to have a heart attack or stroke.

The investigators suspect that patients who get the step count prescriptions will walk more and their arteries will be less hard than the control group. Our study will help find out if this is true. In that case, doctors should take the time to prescribe steps for all their patients with diabetes and/or hypertension.

DETAILED DESCRIPTION:
BACKGROUND: High walking levels reduce myocardial infarction, stroke, and mortality rates in overweight/obese patients with diabetes and/or hypertension, but our own work, led by Nominated Principal Applicant K. Dasgupta, indicates low daily step counts in these patients, at approximately 5,000 steps/day on average with a further 15% reduction during fall and winter. A meta-analysis of physical activity programs indicates that pedometer-based monitoring programs can lead to higher daily step counts, but evidence for impact on arterial health is limited, as is evidence for the effectiveness of a pedometer-based strategy specifically implemented into the usual clinical care of patients with diabetes and/or hypertension. The SMARTER trial will address these knowledge gaps.

PRIMARY RESEARCH QUESTION: Among sedentary overweight/obese adults with diabetes and/or hypertension do physician-delivered step count prescriptions integrated into usual care reduce arterial stiffness more than usual care alone, over a one-year period? Arterial stiffness (primary outcome), a summative indicator of arterial health, is more precise and reliable than individual risk factors. An analysis of the Framingham Heart Study demonstrated that, even after adjustment for traditional risk factors, increased arterial stiffness was independently associated with a 48% increase in vascular disease risk. Co-Principal Applicant S. Daskalopoulou is an expert in the noninvasive assessment of arterial stiffness and has a well-equipped Vascular Lab funded through a CFI grant.

STUDY DESIGN: Randomized, allocation concealed, single-blind (outcome assessors), intervention allocation ratio 1:1, multisite clinical trial. This design will allow for the level A evidence necessary to justify widespread change in clinical practice.

TRIAL SYNOPSIS: Given that the majority of diabetes and hypertension patients are managed in primary care settings, the SMARTER trial interventions will be delivered through the large network of primary care clinics accessible to Co-Principal Applicant E. Rosenberg as well as diabetes and internal medicine clinics throughout Montreal where patients may receive their primary diabetes and hypertension follow-up. Twenty-four collaborating physicians have been identified. Physicians/clinic staff will obtain assent from candidates within their practice for contact by the SMARTER coordinator. The number of collaborating physicians continues to be increased, including physicians at primary care, diabetes, hypertension, internal medicine, and endocrinology clinics. Eligibility: Candidates will be adults with 25≤BMI<40 kg/m2 followed for diabetes and/or hypertension and sedentary to somewhat active. Evaluations: Formal trial evaluations, conducted at baseline and 12 months, will include assessments of arterial stiffness (carotid femoral pulse wave velocity measured noninvasively with applanation tonometry); step counts (pedometer with concealed window) and physical activity (accelerometer) worn for one week; fitness (exercise stress test; ˙VO2max); anthropometric parameters; and individual vascular risk factors. Intervention arm: The physician gives the active trial participants a pedometer, log book, and a step count prescription based on the baseline daily step count. The time frame for a > 3,000 steps/day net increase is 10 months for sedentary participants (<5,000 steps/day), 7 months for low active participants (5,000-7,499 steps/day), and 5 months for somewhat active participants (7,500-9,999 steps/day). There will be four clinic visits over one year. Control arm: Same visit frequency with advice to engage in 30-60 minutes of activity on most days of the week. Sample Size: Allowing for a loss to follow-up of up to 17% based on our previous studies, investigators will require a sample size of 364 individuals (i.e. 182 per arm) to detect a 10% difference in change in arterial stiffness between our active and control arms to an accuracy of +/- 5% over a one-year period. Analysis: Intention-to-treat. Between-arm differences in 'after minus before changes' with 95% CIs for main analysis.

Addedum to stress testing: Due to timeline limitations, we were obliged to forego stress testing assessments as of October 20, 2014. This does not impact our primary outcome. Moreover, stress testing is not required when engaging in a walking program in type 2 diabetes. We will be able to assess impacts of the intervention on fitness (secondary outcome) in a subgroup of patients (i.e., those who completed assessments before October 20, 2014).

IMPORTANCE: With increasing numbers of diabetes and hypertension patients, there is a pressing need for effective and efficient clinical practice strategies to help physicians support their patients to achieve the arterial health benefits of higher physical activity levels. The SMARTER trial seeks to provide such a tool. If effectiveness is demonstrated, all efforts will be made for the inclusion of our approach in Clinical Practice Guidelines for diabetes and hypertension, and investigators will develop training tools (manuals, websites, CD-ROMs) to allow maximal uptake of our proposed strategy.

AN OBSERVATIONAL SUBSTUDY: Novel Real-Time Measurement of Physical Activity Patterns in Type 2 Diabetes and Hypertension Through GPS Monitoring and Accelerometry

In addition to the main clinical trial, we are conducting additional measurements among consenting type 2 diabetes patients in order to examine the effects of the walkability of their home neighbourhood on their baseline step count and time at different physical activity intensities (accelerometer measurement already being performed through SMARTER). The additional measurements include wearing a Geographical Positioning Systems (GPS) device for the 7-day period that they wear the pedometer with concealed viewing window and accelerometer. The GPS device collects time-stamped location information such that X,Y coordinates are collected. These are used to determine the times that they are within or outside neighbourhood buffer zones.

For the assessment of neighbourhood walkability,the parameters assessed include population density, pedestrian-friendly design and diversity of destinations - commonly referred to in the urban planning literature as the 3D's. The variables that best capture density, design, and diversity include residential density, street connectivity and land use mix. Residential density is defined as the number of residences per square kilometre of residential land area. Street connectivity is defined as the number of ≥3-way intersections per square kilometre in neighbourhood, where a greater number of intersections facilitates movement between origins (e.g., residences) and destinations (e.g., shops and parks).Land-use mix is a measure of the number of different land uses located within a neighbourhood.Land use mix is assessed via an entropy score - a value between zero and one that captures the degree of heterogeneity of land uses in a neighbourhood. A subcomponent of land use mix that may be a particularly important for encouraging individuals to walk within their neighbourhood and that is easily incorporated into the design of new neighbourhoods is greenspace/recreational land area.

We are using Geographical Information System (GIS) mapping (computer-based assessment of neighbourhood characteristics derived from existing data sources that have some spatially referenced identification, such as a home address) to measure these facets of neighbourhood walkability.In brief, each of the variables will be derived by geocoding participants six-digit home postal codes, constructing 1-kilometre polygonal buffers zones around each participants home address (i.e., a geographical zone around the centroid of the postal code area) and calculating the measures of interest for each neighbourhood using tools within a GIS software package (ArcGIS) and publically available shape files.

Means and standard deviations will be used to describe the number of steps per day occurring specifically in home neighbourhoods (i.e., as determined through GPS) and overall. Multiple linear regression analyses will be used to assess the relationship between 1) home neighbourhood environments and the number of steps taken per day in the home neighbourhood and 2) home neighbourhood environments and the number of steps taken per day taken in any location. These analyses will be repeated with time at moderate to vigorous activity in lieu of steps as the outcome variable. Several variables measured through SMARTER will be considered for exclusion in models (e.g., age, sex, educational level, BMI).

This observational substudy is partly funded by an operating grant from the Heart and Stroke Foundation (Quebec) awarded to K. Dasgupta (Principal Investigator) and Nancy Ross (Co-Principal Investigator on substudy) and is being led by Samantha Hajna, their doctoral candidate student.

ELIGIBILITY:
Inclusion Criteria:

* Followed by a SMARTER collaborating doctor
* BMI ≥ 25 kg/m2 but < 40 kg/m2 (i.e. overweight to class II obese)
* Type 2 diabetes and/or hypertension
* Conversant in either English or French

Exclusion Criteria:

* ≥ 150 minutes of leisure time physical activity per week be self- report
* Acute or chronic co-morbid conditions that may affect the ability or likelihood to adhere to trial procedures (e.g. inflammatory arthritis, active malignancy, major depression or other significant psychiatric disorders, and/or significant visual impairment)
* Pregnancy/planning a pregnancy
* Baseline step count averaging ≥ 10,000 steps/day at baseline assessment
* Arrhythmia that prevents accurate assessment of carotid-femoral pulse wave velocity (e.g., atrial fibrillation)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change in arterial stiffness | one year
  Arterial stiffness will be assessed at baseline and one year by measurement of carotid femoral pulse wave velocity through applanation tonometry.

SECONDARY OUTCOMES:
change in daily step count | one year
  Step counts will be computed at baseline and final assessments using a Yamax SW-200, based on one week of recording.
change in physical activity | one year
  Change in overall activity will be computed from one week of accelerometry data collected at baseline and at one year
change in physical fitness | one year
  Change in physical fitness will be computed using data collected through maximal exercise stress testing at baseline and one year
weight change from baseline | one year
  Participants will be weighed at baseline and one year in light clothes, without shoes. Change in weight and percentage change in weight from baseline will be computed.
body mass index change from baseline | one year
  Height will be measured using a mounted stadiometer. Body mass index (BMI) will be computed as weight in kg divided by height in meters squared. Change in BMI will be calculated using measurements at baseline and at one year.
change in waist circumference | one year
  Waist circumference will be measured midway between the iliac crest and the lower rib margin. Change in waist circumference will be computed based on data from baseline and one year.
change in waist- to- hip ratio | one year
  Hip circumference will be measured at the point of greatest posterior extension of the buttocks. Waist (in cm) to hip (in cm) ratio (WHR) will be computed and change in WHR will be determined using data from baseline and one year.
change in systolic blood pressure | one year
  The participant will sit at rest for at least five minutes and then undergo blood pressure assessment using the BpTRU Blood Pressure Monitor (seated position, arm supported). The blood pressure assessments will be at two- minute intervals with the patient supine and the measurement in the right arm. The first value will be discarded and the last five measurements averaged.
change in insulin resistance | one year
  Using fasting glucose and fasting insulin measurements, insulin resistance will be computed using the Homeostatic Model Assessment- Insulin Resistance (HOMA- IR) equation [Fasting glucose (mmol/L) X Fasting insulin (mU/L) ÷ 22.5].
change in hemoglobin A1C in diabetes patients | one year
  Change in hemoglobin A1C will be ascertained for diabetes patients between baseline and one year. A1C will be measured with an HPLC analyzer.
change in total cholesterol | one year
  Total cholesterol will be measured using spectrophotometer at baseline and one year
change in high density lipoprotein cholesterol | One year
  High density lipoprotein cholesterol will be measured using spectrophotometer at baseline and one year
Change in triglyceride levels | One year
  Triglyceride levels will be measured using spectrophotometer at baseline and one year
change in low density lipoprotein cholesterol | one year
  The low density lipoprotein cholesterol will be calculated using the Friedewald equation at baseline and one year, based on total cholesterol and high density lipoprotein cholesterol values measured using spectrophotometer.
change in apolipoprotein A1 | one year
  Apolipoprotein A1 will be measured using the turbimetric method at baseline and one year.
change in Apolipoprotein B | One year
  Apolipoprotein B will be measured using the turbimetric method at baseline and one year.
change in Apolipoprotein A1 to B ratio | one year
  Apolipoproteins A1 and B will be measured using the turbimetric method at baseline and one year and the A1 to B ratio computed at these time points
change in total cholesterol to high density lipoprotein cholesterol ratio | one year
  Total cholesterol and high density lipoprotein cholesterol will be measured using spectrophotometer at baseline and at one year; the total cholesterol to high density lipoprotein cholesterol ratio will be computed at both of these time points
change in high sensitivity C-reactive protein | one year
  High sensitivity C-reactive protein will be assayed through an immunonephelometric method at baseline and one year
change in antihypertensive medication use | one year
  Investigators will assess type and dose of antihypertensive medications at baseline and one year and assess whether there has been a net increase, decrease, or no change in medication use.
change in antihyperglycemic medication | one year
  Investigators will assess type and dose of antihyperglycemic medications at baseline and one year and assess whether there has been a net increase, decrease, or no change in medication use.
change in lipid- lowering medications | one year
  Investigators will assess type and dose of lipid- lowering medications at baseline and one year and assess whether there has been a net increase, decrease, or no change in medication use.
change in diastolic blood pressure | one year
  The participant will sit at rest for at least five minutes and then undergo blood pressure assessment using the BpTRU Blood Pressure Monitor (seated position, arm supported). The blood pressure assessments will be at two- minute intervals with the patient supine and the measurement in the right arm. The first value will be discarded and the last five measurements averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MD, MSc, Principal Investigator — McGill University and McGill University Health Centre; Stella Daskalopoulou, MD, PhD, Principal Investigator — McGill University and McGill University Health Centre; Ellen Rosenberg, MD, Principal Investigator — McGill University and St. Mary's Hospital Center
Locations (6):
- Canada (6):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - McGill University Health Centre - Royal Victoria Hosptial, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Lakeshore General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooke AB, Daskalopoulou SS, Dasgupta K. The impact of accelerometer wear location on the relationship between step counts and arterial stiffness in adults treated for hypertension and diabetes. J Sci Med Sport. 2018 Apr;21(4):398-403. doi: 10.1016/j.jsams.2017.08.011. Epub 2017 Aug 24. PMID 28855085
- [Background] Cooke AB, Pace R, Chan D, Rosenberg E, Dasgupta K, Daskalopoulou SS. A qualitative evaluation of a physician-delivered pedometer-based step count prescription strategy with insight from participants and treating physicians. Diabetes Res Clin Pract. 2018 May;139:314-322. doi: 10.1016/j.diabres.2018.03.008. Epub 2018 Mar 10. PMID 29530385
- [Background] Dasgupta K, Rosenberg E, Daskalopoulou SS; SMARTER collaborators. Step Monitoring to improve ARTERial health (SMARTER) through step count prescription in type 2 diabetes and hypertension: trial design and methods. Cardiovasc Diabetol. 2014 Jan 6;13:7. doi: 10.1186/1475-2840-13-7. PMID 24393423
- [Background] Hajna S, Kestens Y, Daskalopoulou SS, Joseph L, Thierry B, Sherman M, Trudeau L, Rabasa-Lhoret R, Meissner L, Bacon SL, Gauvin L, Ross NA, Dasgupta K; Diabetes, GPS, and Walkablilty Study Group. Neighbourhood walkability and home neighbourhood-based physical activity: an observational study of adults with type 2 diabetes. BMC Public Health. 2016 Sep 9;16(1):957. doi: 10.1186/s12889-016-3603-y. PMID 27613233
- [Background] Dasgupta K, Rosenberg E, Joseph L, Cooke AB, Trudeau L, Bacon SL, Chan D, Sherman M, Rabasa-Lhoret R, Daskalopoulou SS; SMARTER Trial Group. Physician step prescription and monitoring to improve ARTERial health (SMARTER): A randomized controlled trial in patients with type 2 diabetes and hypertension. Diabetes Obes Metab. 2017 May;19(5):695-704. doi: 10.1111/dom.12874. Epub 2017 Feb 22. PMID 28074635
- [Background] Dasgupta K, Rosenberg E, Joseph L, Trudeau L, Garfield N, Chan D, Sherman M, Rabasa-Lhoret R, Daskalopoulou SS. Carotid femoral pulse wave velocity in type 2 diabetes and hypertension: capturing arterial health effects of step counts. J Hypertens. 2017 May;35(5):1061-1069. doi: 10.1097/HJH.0000000000001277. PMID 28129250
- See also: BMC Public Health paper — https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-016-3603-y
- See also: Cardiovascular Diabetololy paper — https://cardiab.biomedcentral.com/articles/10.1186/1475-2840-13-7